CLINICAL TRIAL: NCT01678911
Title: Efficacy of Gralise® for Chronic Pelvic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study ended due to difficulties in recruitment and low enrollment.
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Dr. Norman Harden, Director, Center for Pain Studies, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RIC_Dep_CPP_2012
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Irritable Bowel Syndrome; Ulcerative Colitis; Interstitial Cystitis; Prostatitis; Pelvic Pain
Keywords: Pelvic Pain; Chronic Pelvic Pain; Irritable Bowel Syndrome; IBS; Ulcerative Colitis; UC; Interstitial Cystitis; IC; Prostatitis; Pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Colitis, Ulcerative; Cystitis, Interstitial; Prostatitis; Pelvic Pain; Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo then Gralise (Placebo Comparator): Subjects may receive a pill with no medicine (placebo) for phase 1. Subject washout, then cross over to Gralise in Phase 2.
  Interventions: Drug: Gralise
- Gralise then Placebo (Active Comparator): Subjects recieve Gralise (a long acting gabapentinoid) for phase 1.Subject washout, then cross over to placebo in Phase 2.
  Interventions: Drug: Gralise

INTERVENTIONS:
Drug: Gralise — Subjects will start at 600mg and titrate up by 600mg a week for two weeks (to 1800mg), then remain on 1800mg steady state dose of medication (or placebo pills) for 2 weeks. If intolerable side effects occur, the dose may be reduced to last tolerable dose at the discretion of the PI. A 2-week down-titration will be used. Subjects will have 1 week of "wash-out" before repeating the above procedure for the other arm of the study (placebo or medication).
  Other Names: Gabapentin

SUMMARY:
This study is done to investigate the pain relieving effects of the study drug Gralise (a novel long acting gabapentinoid) for people who experience chronic pelvic pain. Subjects with Irritable Bowel Syndrome, Interstitial Cystitis, Ulcerative Colitis, and Prostatitis will be recruited. The purpose of this research is to look at how the study drug can be used to benefit people who experience this type of pain. This is a phase IV study done to study the safety and effectiveness of the drug. At this point the drug has been approved by the Food and Drug Administration and has been reported to be well tolerated and effective in the treatment of various chronic pain conditions, particularly in neuropathic pain. About 36 subjects will take part in this study.

DETAILED DESCRIPTION:
As a participant in this study, you will be asked to come to the Rehabilitation Institute of Chicago (RIC), Center for Pain Studies (446 E Ontario St. Suite 1011, Chicago, IL 60611). Your part in this study will last for 15 weeks and will involve 4 visits to the Rehabilitation Institute of Chicago and anywhere from weekly phone calls to phone calls every other day.

If you are in this study, you will be placed in one of two study groups: one group will receive the study drug followed by a placebo and the second group will receive a placebo followed by the study drug. The amount of weeks on placebo versus the study drug will not be equal. You will be assigned a study group by chance using a process similar to the flip of a coin. This process is called randomization. Neither you nor the study staff will select the group you will be in. However, if you have a medical emergency, we can get this information. A placebo looks like the study drug but is an inactive substance that has no medication. Researchers use a placebo to see if the study drug works better or is safer than not taking anything.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* English speaking
* able to give consent
* willing to use electronic diary during entire length of the study
* has 'chronic' pelvic pain
* Meets one of the following diagnostic criteria for one of the following: Irritable Bowel Syndrome (IBS) Ulcerative Colitis (UC), Interstitial Cystitis (IC), and Prostatitis

Exclusion Criteria:

* allergic to gabapentin or inactive ingredients
* taking gabapentinoids (i.e. gabapentin or pre-gabalin)
* with severe or unmanaged psychiatric disturbance (at PI discretion)
* with severe ongoing or unaddressed medical conditions (esp. Renal or Hepatic disease, uncontrolled hypertension), rheumatologic disease, narrow angle glaucoma, hyponatremia, clotting disorders, uncontrolled seizure disorder or urinary retention.
* who plan to change their therapeutic regimen during the course of the trial (e.g. start physical therapy, massage, medications, injections, etc.)
* with acute pain

Female subjects:

* pregnant or plan to become pregnant
* gave birth within the last 6 months
* breastfeeding
* episodic visceral pain (e.g. endometriosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Harden, MD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute Of Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: Site Contact Info — http://www.ric.org/research/centers/pain/index.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 Subjects enrolled in the study and started a single-blind placebo lead-in period. Of those, 5 were randomized. 6 subjects did not continue and were either lost to follow-up, chose not to continue, or exhibited a large placebo response and no longer met the criteria to continue in the study.
Groups:
- Placebo, Then Gralise: Subjects may receive a pill with no medicine.
- Gralise Then Placebo: Gralise (a long acting gabapentinoid)
  Gralise: Subjects will start at 600mg and titrate up by 600mg a week for two weeks (to 1800mg), then remain on 1800mg steady state dose of medication (or placebo pills) for 2 weeks. If intolerable side effects occur, the dose may be reduced to last tolerable dose at the discretion of the PI. A 2-week down-titration will be used. Subjects will have 1 week of "wash-out" before repeating the above procedure for the other arm of the study (placebo or medication).
Period: First Intervention
Arm/Group | Placebo, Then Gralise | Gralise Then Placebo
Started | 4 | 1
Cross Over | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo, Then Gralise | Gralise Then Placebo
Started | 4 | 1
Completed | 2 | 1
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All randomized subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: McGill Pain Questionnaire - Short Form
Description: The MPQ-SF is a well-validated pain measure that permits separation of the sensory and affective components of pain, which are averaged to compute a total score. The scale ranges from 0-10 (0=no pain, 10=the most pain).
Time Frame: 4 Visits over a 15 week period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Then Gralise | Gralise Then Placebo
Number analyzed (Participants) | 4 | 1
units on a scale
  change from baseline after intervention 1 | -0.34 (1.78) | .04 (0)
  change from baseline after intervention 2 | 1.05 (0.45) | .41 (0)

2. Secondary Outcome: Pain Anxiety Symptoms Scale
Description: The Pain Anxiety Symptoms Scale (PASS) is an anxiety scale from 0 - 100, where 0 = no anxiety and 100 = the most anxiety.
Time Frame: 4 Visits over an 8 week period
Measure: Mean (Standard Deviation); unit: units on the PASS scale
Arm/Group | Placebo Then Gralise | Gralise Then Placebo
Number analyzed (Participants) | 4 | 1
units on the PASS scale
  mean change after intervention 1 | -5.8 (18.0) | -4 (0)
  mean change after intervention 2 | 9.0 (22.6) | -5 (0)

3. Secondary Outcome: Pain Disability Index
Description: The PDI is a seven-item, validated instrument that assesses perceived disability in seven key life areas. It provides a total disability score, and is an indirect measure of self efficacy. The Pain Disability Scale is a scale from 0 - 70, where 0 = no Disability and 70 = the most Disability.
Time Frame: 4 visits over an 8 week period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Then Gralise | Gralise Then Placebo
Number analyzed (Participants) | 4 | 1
units on a scale
  change after intervention 1 | 4.8 (13.9) | 10 (0)
  change after intervention 2 | 19 (4.2) | 14 (0)

4. Secondary Outcome: Center for Epidemiologic Studies Depression Scale
Description: The CES-D 10 is a 10-item questionnaire that has been validated for the assessment of depressive symptomatology. The Depression Scale is a scale with a sum score from 0 - 30, where 0 = no Depression and 30 = the most Depression.
Time Frame: 4 visits over 15 week period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Then Gralise | Gralise Then Placebo
Number analyzed (Participants) | 4 | 1
units on a scale
  change after intervention 1 | 4.5 (5.7) | -1 (0)
  change after intervention 2 | 7 (2.8) | 0 (0)

5. Secondary Outcome: Patient Global Impression of Change
Description: Patient Global Impression of Change is a self-report questionnaire on which patient indicate their perceived impression of change since the start of the study given the following options: Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse, or Very much Worse.
Time Frame: 4 Visits over 15 weeks
Measure: Number; unit: participants
Arm/Group | Placebo Then Gralise | Gralise Then Placebo
Number analyzed (Participants) | 4 | 1
participants
  improved after intervention 1 | 3 | 0
  no change after intervention 1 | 0 | 1
  worse after intervention 1 | 1 | 0
  improved after intervention 2 | 1 | 0
  no change after intervention 2 | 1 | 0
  worse after intervention 2 | 0 | 1

ADVERSE EVENTS:
Groups:
- Sugar Pill: Subjects may receive a pill with no medicine.
- Gralise: Gralise (a long acting gabapentinoid)
  Gralise: Subjects will start at 600mg and titrate up by 600mg a week for two weeks (to 1800mg), then remain on 1800mg steady state dose of medication (or placebo pills) for 2 weeks. If intolerable side effects occur, the dose may be reduced to last tolerable dose at the discretion of the PI. A 2-week down-titration will be used. Subjects will have 1 week of "wash-out" before repeating the above procedure for the other arm of the study (placebo or medication).
Arm/Group | Sugar Pill | Gralise
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill (N=5) | Gralise (N=5)
Drowsiness (General disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
This study was terminated early due to low recruitment. Therefore, the data presented represents a very small sample, with low 'n's in each group. The data tables represent all available data for the small sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No